CLINICAL TRIAL: NCT06959043
Title: Therapeutic Strategies for Type 2 Diabetes Based on Lifestyle Changes: Plant-based Diet and Physical Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Elizabeth Rossi da Silva (Other)
Collaborators: Clínica e Spa Vida Natural (Unknown); Probiotical Spa (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Maria Elizabeth Rossi da Silva, MD, PhD, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cappesq
Record Dates: First submitted 2025-03-09; First posted 2025-05-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Insulin Resistance; Inflamation; Gut Microbiomes
Keywords: Type 2 Diabetes Mellitus; Insulin Resistance; Inflamation; Metabolic Syndrome; Physical Exercise; Gut Microbiome; Plant-based Diet; Lifestyle Interventions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Metabolic Syndrome; Motor Activity | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, randomized clinical trial. Patients will be informed about the type of therapy they will receive at the clinic, which includes a strict vegetarian diet and regular physical exercises, as well as the importance of adhering strictly to the prescribed instructions.
  A total of 60 patients will be recruited, with a maximum of six participants per four-week cycle. They will be randomized and allocated to the following treatment groups:
  Group 1: Strict vegetarian diet (SVD) + regular physical exercise (RPE) (n=30). Group 2: SVD + RPE + administration of a probiotic pool (n=30).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strict Vegetarian Diet, Regular Physical Exercise, and Placebo Administration (Placebo Comparator): Participants in this group will follow a strict vegetarian diet (SVD) combined with regular physical exercise (RPE) for four weeks. The diet will consist of plant-based foods rich in fiber and bioactive compounds, with a controlled macronutrient distribution. Physical activity will include structured aerobic and resistance exercises supervised by a physical educator. Instead of probiotic supplementation, participants will receive a placebo administered in the same manner as the probiotic group to ensure blinding.
  Interventions: Dietary Supplement: Placebo Administration
- Strict Vegetarian Diet, Regular Physical Exercise, and Probiotic Supplementation (Experimental): Participants in this group will receive the same strict vegetarian diet (SVD) and regular physical exercise (RPE) as Arm 1. In addition, they will take a probiotic supplement containing a combination of four different strains, administered twice daily for four weeks. This group aims to assess the potential additional metabolic benefits of probiotic supplementation in individuals with type 2 diabetes.
  Interventions: Dietary Supplement: Probiotic Supplementation

INTERVENTIONS:
Dietary Supplement: Probiotic Supplementation — Participants will follow the same strict vegetarian diet and regular physical exercise as in Intervention 1. Additionally, they will receive a probiotic supplement, taken twice daily for four weeks. This aims to evaluate the metabolic impact of probiotics in type 2 diabetes.
  Other Names: Probiotic
  Arms: Strict Vegetarian Diet, Regular Physical Exercise, and Probiotic Supplementation
Dietary Supplement: Placebo Administration — Participants will follow a strictly plant-based diet rich in fiber and bioactive compounds, with controlled macronutrient distribution. Regular physical exercise includes supervised aerobic and resistance training sessions. The intervention lasts four weeks. Instead of probiotic supplementation, participants will receive a placebo, administered in the same manner as the probiotic group to maintain blinding.
  Other Names: Placebo
  Arms: Strict Vegetarian Diet, Regular Physical Exercise, and Placebo Administration

SUMMARY:
The study evaluates the impact of a strict vegetarian diet combined with regular physical exercise and the use of probiotics on metabolic, inflammatory, and epigenetic parameters in patients with type 2 diabetes. It aims to determine the influence of these interventions on gut microbiota, glycemic control, body composition, insulin resistance, and quality of life.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effects of a strict vegetarian diet (SVD) combined with regular physical exercise (RPE), with or without probiotic supplementation, on key metabolic and physiological parameters in patients with type 2 diabetes mellitus (T2DM). Participants will be monitored for changes in glycemic control, insulin resistance (IR), liver function (elastography and ultrasound), metabolomic profile, muscle composition (biopsy), cholesterol efflux, and gene expression.

Glycemic Control Glycemic control will be assessed through glycated hemoglobin (HbA1c), fasting glucose, fructosamine, and oral meal tolerance test (OMTT). A standardized dietary test (500 kcal plant-based meal) will be conducted at baseline and post-intervention, measuring postprandial glucose, insulin, proinsulin, C-peptide, and incretin hormones (GLP-1, GIP).

Insulin Resistance (IR) IR will be evaluated using HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) and fasting insulin levels. The study will also analyze inflammatory markers (TNF-α, IL-1β, IL-6, IFN-γ), as chronic low-grade inflammation plays a crucial role in IR development.

Elastography and Ultrasound (US) Liver ultrasound and transient elastography (FibroScan®) will be performed to assess hepatic steatosis and fibrosis, which are highly prevalent in T2DM. The effects of dietary and probiotic interventions on liver fat content, liver stiffness, and metabolic liver function will be analyzed.

Metabolome Analysis Metabolomic profiling will be conducted through mass spectrometry-based analysis of fasting and postprandial plasma samples. The study will evaluate amino acids, lipids, short-chain fatty acids, bile acids, ketone bodies, and glycolysis-related metabolites to understand how dietary and microbiome changes influence metabolic pathways in T2DM.

Muscle Biopsy A vastus lateralis muscle biopsy will be performed in a subgroup of participants (n=24). Samples will be analyzed for fiber composition, extracellular matrix remodeling, mitochondrial function, and inflammatory markers. The role of microRNAs (miR-29a, miR-29b, miR-1, miR-133a/b, miR-206) in muscle insulin sensitivity will also be investigated.

Cholesterol Efflux HDL functionality will be assessed by measuring cholesterol efflux capacity from macrophages exposed to participants' serum. This analysis will provide insight to cardiovascular risk modulation by diet and probiotics in T2DM.

Gene Expression Analysis Peripheral blood lymphocytes will be analyzed for expression of inflammation-related genes (TNF-α, IL-6, IL-1β, IFN-γ, TLR4, TLR5) and longevity-related genes (SIRT1, FOXO1, PGC-1α, P53). These markers will help determine how dietary and probiotic interventions influence immune response, cellular aging, and metabolic regulation.

Microbiota analysis This study will assess how a strict vegetarian diet and probiotic supplementation influence gut microbiota composition and functionality in individuals with T2DM. Stool samples will be collected before and after the intervention (4 weeks) and analyzed using 16S rRNA sequencing (NGS platforms: Ion Torrent PGM or Illumina MiSeq).

Microbiota diversity (alpha and beta diversity metrics) and the relative abundance of key bacterial taxa (Bacteroides, Firmicutes, Akkermansia, Prevotella, Bifidobacterium, Lactobacillus) will be evaluated. Functional analysis will include metagenomic predictions (PICRUSt2), short-chain fatty acid (SCFA) production, and microbial metabolic pathways.

The impact of probiotic supplementation (B. breve BR03, B. breve B632, B. longum 04, L. reuteri LRE11) will be assessed by comparing gut microbiota changes between the probiotic and placebo groups, focusing on butyrate-producing bacteria, lactate-utilizing species, and intestinal barrier integrity markers.

The intervention will last four weeks, followed by 12 months of telemedicine follow-up. This study aims to provide new insights into the role of lifestyle interventions in metabolic regulation, inflammation, and gut microbiota modulation in T2DM, potentially offering novel therapeutic strategies beyond pharmacological approaches.

ELIGIBILITY:
Inclusion Criteria:

* Have a medical diagnosis of type 2 diabetes for a maximum of 5 years.
* Be omnivorous; Have a Body Mass Index (BMI) ≥ 25 kg/m2 and < 40 kg/m2;
* Be between the ages of 45 and 70, both genders.
* Women should be in the postmenopausal stage;
* Use no more than three hypoglycemic medications in total;
* Have the availability for a four-week consecutive hospitalization at CSVN.

Exclusion Criteria:

* Be using insulin, anti-obesity medications, antibiotics, and/or probiotic supplements in the 2 months preceding data collection;
* Use of alcohol or tobacco;
* Have limited mobility and a previous diagnosis of cardiopulmonary diseases;
* Report current or previous (within the past two months) diarrhea during screening;
* Have liver or kidney failure and uncontrolled endocrine disorders (hypothyroidism, hypogonadism, and adrenal insufficiency);
* Have eating disorders or have undergone bariatric surgery.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 4 weeks post-intervention
  Body mass index (BMI) will be calculated from height and weight (weight in kg / height in m²) to assess the impact of the intervention on overall body weight regulation. This outcome reflects metabolic improvement and lifestyle adherence.
  Unit of Measure: kg/m²
Change in Waist, Abdominal, and Hip Circumference | Baseline and 4 weeks post-intervention
  Waist, abdominal, and hip circumferences will be measured using a standardized flexible tape method. These anthropometric parameters are indicators of central fat distribution and associated cardiometabolic risk. Measurements will follow WHO recommendations.
  Unit of Measure: cm
Change in Waist-to-Hip Ratio (WHR) | Baseline and 4 weeks post-intervention
  Waist-to-hip ratio (WHR) will be calculated by dividing waist circumference by hip circumference. This index is used to evaluate body fat distribution and the risk of metabolic disorders, particularly central obesity, in individuals with T2DM.
  Unit of Measure: Ratio (unitless)
Change in Functional Aerobic Capacity (1-Mile Walk Test) | Baseline and 4 weeks post-intervention
  Aerobic capacity will be assessed using the 1-Mile Walk Test. Participants will be instructed to walk one mile as fast as possible on a flat surface, and the time to completion will be recorded. The objective is to evaluate improvements in cardiovascular endurance following the intervention.
  Unit of Measure: Time in minutes
Change in Functional Mobility (Up and Go Test) | Baseline and 4 weeks post-intervention
  Functional mobility will be assessed using the "Up and Go" test. Participants will be timed as they rise from a seated position, walk three meters, turn around, walk back to the chair, and sit down. The test is used to detect improvements in balance, mobility, and lower-limb function in response to the intervention.
  Unit of Measure: Time in seconds
Change in Fasting Blood Glucose | Baseline and 4 weeks post-intervention
  Fasting plasma glucose will be measured after 8-12 hours of fasting by glucose-oxidase method to evaluate improvements in basal glycemic levels.
  The goal is to determine whether the intervention improves glucose homeostasis in patients with T2DM.
  Unit of Measure: mg/dL
Change in Postprandial Glucose Levels | Baseline and 4 weeks post-intervention
  Two-hour postprandial glucose will be measured using capillary or venous blood samples by glucose-oxidase method after a standardized meal. The goal is to evaluate improvements in glycemic response to food intake due to the intervention.
  Unit of Measure: mg/dL
Change in Glycated Hemoglobin (HbA1c) | Baseline and 4 weeks post-intervention
  Glycated hemoglobin (HbA1c) levels will be measured in venous blood samples using HPLC to assess long-term glycemic control. The main hypothesis is that the combined intervention of a plant-based diet, physical exercise, and probiotics will significantly reduce HbA1c levels compared to baseline.
  Unit of Measure: % HbA1c

SECONDARY OUTCOMES:
Change in Liver Enzymes (AST, ALT, GGT) | Baseline and 4 weeks post-intervention
  Serum levels of liver enzymes (AST, ALT, GGT) will be measured using automated enzymatic assays to evaluate liver function and detect possible hepatocellular injury or metabolic improvements after the intervention.
  Unit of Measure: U/L
Change in Standard Lipid Profile | Baseline and 4 weeks post-intervention
  Serum levels of total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides will be measured by enzymatic colorimetric assays. These parameters are essential for assessing cardiometabolic risk in patients with T2DM.
  Unit of Measure: mg/dL
HDL Function and Lipid Profile | Baseline and 4 weeks post-intervention
  HDL function will be evaluated by measuring cholesterol efflux capacity in vitro using labeled macrophage assays. The result reflects HDL's ability to remove cholesterol from peripheral tissues, a key anti-atherogenic property.
  Unit of Measure: % cholesterol efflux
Change in C-Reactive Protein (CRP) Levels | Baseline and 4 weeks post-intervention
  C-reactive protein (CRP), a marker of systemic low-grade inflammation and cardiovascular risk, will be measured in plasma using high-sensitivity Luminex assay.
  Unit of Measure: mg/L
Change in Plasma Cytokine Levels | Baseline and 4 weeks post-intervention
  Plasma concentrations of proinflammatory cytokines TNF-α, IL-6, IL-1β, and IFN-γ will be measured using the Luminex multiplex assay. These markers are associated with systemic inflammation and insulin resistance in patients with T2DM.
  Unit of Measure: pg/mL
Metabolomic and Biochemical Markers | Baseline and 4 weeks post-intervention
  Metabolomic profiling will assess amino acids, fatty acids, and glucose/lipid-related metabolites in plasma using mass spectrometry. Both fasting and postprandial samples will be analyzed.
  Unit of Measure: μmol/L
Change in expression of Metabolism- and Inflammation-Related microRNAs | Baseline and 4 weeks post-intervention
  Expression levels of specific microRNAs involved in metabolic and inflammatory pathways will be measured in plasma and tissue samples by qPCR.
  Unit of Measure: Fold change
Change in Expression of Inflammatory Genes | Baseline and 4 weeks post-intervention
  Gene expression of inflammatory markers will be analyzed in peripheral blood lymphocytes using NGS.
  Unit of Measure: Fold change
Change in Inflammatory Gene Expression in Lymphocytes and Skeletal Muscle | Baseline and 4 weeks post-intervention
  Expression of genes encoding inflammatory mediators will be assessed by RT-qPCR in samples from peripheral blood lymphocytes and skeletal muscle. Expression will be reported as fold change compared to baseline.
  Unit of Measure: Fold change
Change in Fasting Insulin, Proinsulin, and C-Peptide Levels | Baseline and 4 weeks post-intervention
  Fasting serum levels of insulin, proinsulin, and C-peptide will be measured using specific immunoassays. These markers collectively provide information about pancreatic β-cell function, insulin secretion, and metabolic status in patients with T2DM. Measurements will assess the effect of the intervention on pancreatic hormone production and secretion.
  Unit of Measure: ng/mL
Change in Insulin Resistance Assessed by HOMA-IR | Baseline and 4 weeks post-intervention
  Insulin resistance will be evaluated using the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting glucose and insulin concentrations. Higher HOMA-IR values indicate greater insulin resistance.
  Unit of Measure: Index value (unitless)
Change in Incretin Hormone Levels (GLP-1 and GIP) | Baseline and 4 weeks post-intervention
  Fasting plasma levels of the incretin hormones GLP-1 and GIP will be assessed using ELISA assays. These hormones play essential roles in glucose homeostasis by enhancing insulin secretion.
  Unit of Measure: pmol/L
Changes in Gut Microbiota Composition | Baseline and 4 weeks post-intervention
  Microbial composition will be analyzed by 16S rRNA sequencing of fecal samples. Outcomes include alpha- and beta-diversity indices and the relative abundance (%) of specific bacterial taxa. These analyses aim to assess the impact of the dietary and probiotic intervention on gut microbiota in T2DM patients.
  Unit of Measure: Diversity index, % abundance
Change in Liver Steatosis Assessed by Abdominal Ultrasound | Baseline and 4 weeks post-intervention
  Hepatic steatosis will be assessed using abdominal ultrasound performed by trained radiologists. Ultrasound evaluation will classify the degree of steatosis based on echogenicity criteria (mild, moderate, or severe). The purpose is to monitor the presence and severity of hepatic fat infiltration among participants with T2DM and to evaluate their response to the intervention.
  Unit of Measure: Steatosis grade (mild, moderate, severe)
Change in Liver Fat and Fibrosis Assessed by Transient Elastography | Baseline and 4 weeks post-intervention
  Hepatic fat content and liver stiffness will be evaluated by transient elastography (FibroScan) to assess changes in hepatic steatosis and fibrosis after the intervention. Measurements will be expressed in kilopascals (kPa).
  Unit of Measure: kPa
Change in Depressive Symptoms Measured by the Beck Depression Inventory - Second Edition (BDI-II) | Baseline and 12 weeks post-intervention
  Depressive symptoms will be assessed using the Beck Depression Inventory - Second Edition (BDI-II), a 21-item self-report questionnaire. Each item is scored from 0 to 3, resulting in a total score ranging from 0 to 63. Higher scores indicate greater severity of depressive symptoms. Interpretation of the total score is as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
  Unit of Measure: Total BDI-II score (range: 0-63; higher scores indicate worse outcomes)
Change in Diabetes-Specific Quality of Life Measured by the Diabetes Quality of Life Measure (DQOL) | Baseline and 12 weeks post-intervention
  Diabetes-specific quality of life will be assessed using the Diabetes Quality of Life Measure (DQOL), Brazilian version. The instrument contains 44 items divided into four domains: satisfaction, impact, social/vocational concerns, and diabetes-related concerns. Each item is rated on a 5-point Likert scale. The mean score ranges from 1 to 5, with higher scores indicating worse quality of life. Interpretation of the scores is as follows:
  * 1.0 to 2.0: Very good diabetes-related quality of life
  * 2.1 to 3.0: Moderate quality of life
  * 3.1 to 4.0: Poor quality of life
  * 4.1 to 5.0: Very poor quality of life Unit of Measure: Mean DQOL - Brazil score (range: 1-5; higher scores indicate worse outcomes)
Change in General Well-Being Measured by the Q8RN Questionnaire | Baseline and 12 weeks post-intervention
  General well-being will be assessed using the Q8RN Questionnaire (Eight Natural Remedies Questionnaire), which evaluates eight dimensions of healthy lifestyle habits: nutrition, exercise, water intake, sunlight exposure, temperance, fresh air, rest, and trust in God. Each dimension is assessed through Likert-scale questions, generally rated from 0 to 4 or from 1 to 5, depending on the version. Participants indicate how frequently they engage in each behavior (e.g., "never," "rarely," "sometimes," "often," "always").
  Scores for each dimension can be analyzed separately or summed into a global score. Interpretation: higher scores indicate better adherence to healthy lifestyle practices. The Q8RN results can be used to identify lifestyle areas needing improvement or to track changes over time following educational or health-promotion interventions.
  Unit of Measure: Total Q8RN score (range: 8-40; higher scores indicate better outcomes)
Change in Fasting Glucose During Telemedicine Follow-Up | Every 3 months over a 12-month follow-up period after the intervention
  Fasting plasma glucose will be measured at each telemedicine follow-up visit (every 3 months) over one year to monitor glycemic control. Blood samples will be collected after at least 8 hours of fasting. The intervention aims to improve and maintain fasting glucose levels within target ranges for patients with T2DM.
  Unit of Measure: mg/dL
Change in HbA1c Levels During Telemedicine Follow-Up | Every 3 months over a 12-month follow-up period after the intervention
  HbA1c will be measured at each telemedicine follow-up to evaluate long-term glycemic control. Blood samples will be analyzed to determine the average blood glucose concentration over the preceding 2-3 months. The intervention aims to reduce and stabilize HbA1c levels.
  Unit of Measure: % HbA1c
Change in Lipid Profile During Telemedicine Follow-Up | Every 3 months over a 12-month follow-up period after the intervention
  Serum lipid profile, including total cholesterol, LDL, HDL, and triglycerides, will be assessed at each telemedicine follow-up to monitor cardiometabolic health. These parameters reflect lipid metabolism and cardiovascular risk among patients with T2DM.
  Unit of Measure: mg/dL
Change in Liver Enzymes During Telemedicine Follow-Up | Every 3 months over a 12-month follow-up period after the intervention
  Liver function will be monitored through serum levels of liver enzymes (AST, ALT, and GGT) measured every 3 months. This monitoring helps detect potential hepatic changes and the effect of the intervention on liver health.
  Unit of Measure: U/L

CONTACTS AND LOCATIONS:
Overall Officials: Maria E. R. Silva, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade de São Paulo (USP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The IPD will be available at the end of the study
Access Criteria: The information will be available with reazonable request

REFERENCES:
- [Background] Guasch-Ferre M, Hruby A, Toledo E, Clish CB, Martinez-Gonzalez MA, Salas-Salvado J, Hu FB. Metabolomics in Prediabetes and Diabetes: A Systematic Review and Meta-analysis. Diabetes Care. 2016 May;39(5):833-46. doi: 10.2337/dc15-2251. PMID 27208380
- [Background] Nikiforova VJ, Giesbertz P, Wiemer J, Bethan B, Looser R, Liebenberg V, Ruiz Noppinger P, Daniel H, Rein D. Glyoxylate, a new marker metabolite of type 2 diabetes. J Diabetes Res. 2014;2014:685204. doi: 10.1155/2014/685204. Epub 2014 Nov 27. PMID 25525609
- [Background] Koutnikova H, Genser B, Monteiro-Sepulveda M, Faurie JM, Rizkalla S, Schrezenmeir J, Clement K. Impact of bacterial probiotics on obesity, diabetes and non-alcoholic fatty liver disease related variables: a systematic review and meta-analysis of randomised controlled trials. BMJ Open. 2019 Mar 30;9(3):e017995. doi: 10.1136/bmjopen-2017-017995. PMID 30928918
- [Background] Miraghajani M, Dehsoukhteh SS, Rafie N, Hamedani SG, Sabihi S, Ghiasvand R. Potential mechanisms linking probiotics to diabetes: a narrative review of the literature. Sao Paulo Med J. 2017 Mar-Apr;135(2):169-178. doi: 10.1590/1516-3180.2016.0311271216. PMID 28538869
- [Background] Heppner KM, Perez-Tilve D. GLP-1 based therapeutics: simultaneously combating T2DM and obesity. Front Neurosci. 2015 Mar 20;9:92. doi: 10.3389/fnins.2015.00092. eCollection 2015. PMID 25852463
- [Background] Firouzi S, Majid HA, Ismail A, Kamaruddin NA, Barakatun-Nisak MY. Effect of multi-strain probiotics (multi-strain microbial cell preparation) on glycemic control and other diabetes-related outcomes in people with type 2 diabetes: a randomized controlled trial. Eur J Nutr. 2017 Jun;56(4):1535-1550. doi: 10.1007/s00394-016-1199-8. Epub 2016 Mar 17. PMID 26988693
- [Background] Hopper I, Billah B, Skiba M, Krum H. Prevention of diabetes and reduction in major cardiovascular events in studies of subjects with prediabetes: meta-analysis of randomised controlled clinical trials. Eur J Cardiovasc Prev Rehabil. 2011 Dec;18(6):813-23. doi: 10.1177/1741826711421687. Epub 2011 Aug 30. PMID 21878448
- [Background] Jardine MA, Kahleova H, Levin SM, Ali Z, Trapp CB, Barnard ND. Perspective: Plant-Based Eating Pattern for Type 2 Diabetes Prevention and Treatment: Efficacy, Mechanisms, and Practical Considerations. Adv Nutr. 2021 Dec 1;12(6):2045-2055. doi: 10.1093/advances/nmab063. PMID 34113961
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Barnard ND, Katcher HI, Jenkins DJ, Cohen J, Turner-McGrievy G. Vegetarian and vegan diets in type 2 diabetes management. Nutr Rev. 2009 May;67(5):255-63. doi: 10.1111/j.1753-4887.2009.00198.x. PMID 19386029
- See also: The article reviews molecular mechanisms linking obesity to insulin resistance and highlights the role of physical exercise in reducing inflammation, improving insulin signaling, and contributing to better metabolic control and overall health. — https://pesquisa.bvsalud.org/portal/resource/pt/lil-733971